CLINICAL TRIAL: NCT05208749
Title: A Randomized Controlled Trial Comparing Rates of Peri-procedural Myocardial Infarction After Intravascular Ultrasound and Rotational Atherectomy in Patients With Calcified Coronary Artery Lesions
Brief Title: ShOckwave ballooN or Atherectomy With Rotablation in Calcified Coronary Artery Lesions, the SONAR Trial
Acronym: SONAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Ziekenhuis Oost-Limburg (Other); University Hospital, Ghent (Other); Universitair Ziekenhuis Brussel (Other); Ziekenhuis Netwerk Antwerpen (ZNA) (Other); Imelda Hospital, Bonheiden (Other); AZ Sint-Lucas Brugge (Other); Centre Hospitalier Universitaire Saint Pierre (Other); Hôpital Jolimont (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: S64676
Record Dates: First submitted 2021-12-08; First posted 2022-01-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Calcified Atheroma; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rotablation (Active Comparator): Use of rotational atherectomy first-line if NC balloon does not fully open
  Interventions: Device: Rotablation of shockwave
- Shockwave IVL (Active Comparator): Use of Shockwave IVLS first-line if NC balloon does not fully open
  Interventions: Device: Rotablation of shockwave

INTERVENTIONS:
Device: Rotablation of shockwave — Patients will be randomized to treatment with rotablation or shockwave

SUMMARY:
Percutaneous coronary interventions (PCI) is intended to relieve myocardial ischemia by improving blood flow in the epicardial coronary arteries. However, the efficacy of PCI may be compromised by incidental microvascular obstruction and peri-procedural myocardial infarction (PPMI), which occurs in about 10-15% of cases and is associated with increased rates of major adverse cardiovascular events (MACE). The mechanism of PPMI is thought to be related to side branch occlusion, coronary artery dissection and acute microvascular damage caused by embolization of plaque debris during the PCI and is more frequently seen in calcified coronary artery disease. Calcium modification by rotational atherectomy (RA) results in peri-procedural myocardial infarction in 24% of cases and myocardial injury in 70% of cases. The Shockwave coronary intravascular lithotripsy (IVL) balloon catheter emits sonic pressure waves in a circumferential field causing the selective fracture of calcium, altering vessel compliance and permitting further expansion of the vessel wall. This provides a potentially safer alternative to other calcium-modifying devices since there is a low risk of dissection and perforation. It is also proposed that this IVL device reduces the risk of atheromatous embolization, which would reduce the risk of PPMI and microvascular dysfunction. The SONAR Trial is a pilot study measuring peri-procedural myocardial injury, PPMI and microvascular dysfunction in patients (with calcified coronary artery lesions not responding to usual balloon dilatation) randomized to RA or Shockwave IVL. The primary outcome is peri-procedural myocardial infarction. Secondary outcomes include peri-procedural myocardial injury, acute microvascular dysfunction, procedural success, and procedural costs.

DETAILED DESCRIPTION:
In this multicentre, prospective, randomized-controlled open label pilot study the investigators will measure rates of peri-procedural myocardial infarction and changes in microvascular function after PCI in 170 patients (85 per arm) treated with Shockwave intravascular lithotripsy (IVL) versus RA. Patients with moderately and/or severely calcified coronary lesions, which are equally suitable for IVL and RA and do not dilate fully (100%) with an appropriately sized non-compliant balloon at 16 atmospheres, will be recruited. The calcified lesion must be suitable for both IVL and RA and the operator believes that either IVL or RA could be used. The primary outcome will be difference in the rate of peri-procedural myocardial infarction (Type 4a of the universal Definition of Myocardial Infarction). Peri-procedural myocardial injury and infarction will be defined by an increase in high-sensitivity Troponin T according to the Fourth Universal Definition of Myocardial Infarction,15 while microvascular dysfunction will be defined by an Index of Microcirculatory Resistance (IMR) of ≥25.16 Patients will undergo study-related clinical follow up at 30 days and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years.
* The subject has stable or unstable angina pectoris, or a positive functional study for ischemia.
* The subject is eligible for PCI.
* The subject gives consent prior to study inclusion.
* The subject has a calcified lesion that does not dilated fully after balloon angioplasty at 16atm with a ≥2.5mm non-compliant balloon.
* The calcified lesion has a 50-90% diameter stenosis by angiographic assessment.

Exclusion Criteria:

* Previous and/or planned brachytherapy of target vessel.
* Pregnant and/or breast-feeding females or females who intend to become pregnant.
* Patients who intend to have a major surgical intervention within 6 months of enrolment in the study.
* Patients who previously participated in this study.
* Subject has experienced an acute myocardial infarction 72 hours prior to the index procedure, as defined either by the presence of a new Q-wave in 2 or more contiguous leads, or by a CK greater than two times site upper reference limit (URL) with presence of CK-MB greater than the site URL.
* The subject has suffered a stroke or transient ischemic neurological attack or cerebrovascular accident within the past six months, or has any known intracranial mass, arteriovenous malformation, aneurysm or other intracranial pathology.
* The subject has experienced a significant gastrointestinal or genitourinary bleed within the past six months, or has had any active bleeding within two months.
* Planned revascularization of target vessel within 1 year after index procedure.
* Lesions not ideal for Shockwave treatment:
* Longer than 40mm.
* The target vessel contains intraluminal thrombus.
* The subject has had a prior stent in the target lesion, including a 5mm zone proximal and distal to the lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Difference in peri-procedural myocardial infarction (Type 4a) | within 24 hours of index PCI
  Measurements of HS Troponine T at 8hrs, 16hrs and 24 hrs post PCI

SECONDARY OUTCOMES:
Procedural differences (technical and procedural success, procedural characteristics and costs). | periprocedural
  procedural characteristics
Difference in change in IMR between the two groups. | periprocedural
  measurement of IMR before and after PCI
Clinical outcomes at 30-days and 1 year. | 1 year
  clinical outcomes (Major adverse clinical events, including MI, TLR and cardiac death)
IMR change post-PCI in calcified lesions | periprocedural
  measurement of IMR before and after PCI
Peri-procedural myocardial injury incidence | periprocedural
  Measurements of HS Troponine T at 8hrs, 16hrs and 24 hrs post PCI

CONTACTS AND LOCATIONS:
Locations (1):
- University Hopsitals Leuven, Leuven, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No